CLINICAL TRIAL: NCT06361888
Title: A Multicenter, Randomized, Open-label, Active-controlled, Phase II/III Trial to Evaluate the Efficacy and Safety of Surufatinib Combined With Camrelizumab, Nab-paclitaxel, and Gemcitabine Versus Nab-paclitaxel Plus Gemcitabine as the First-line Treatment in Metastatic Pancreatic Cancer
Brief Title: A Phase II/III Trial to Evaluate the Efficacy and Safety of Surufatinib Combined With Camrelizumab, Nab-paclitaxel, and Gemcitabine in Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-012-00CH1
Record Dates: First submitted 2024-03-26; First posted 2024-04-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: First-line treatment in patients
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — camrelizumab; 130-nm albumin-bound paclitaxel; Gemcitabine; surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surufatinib Combined With Camrelizumab, Nab-paclitaxel, and Gemcitabine (Experimental)
  Interventions: Drug: Surufatinib Combined With Camrelizumab, Nab-paclitaxel, and Gemcitabine
- Nab-paclitaxel Plus Gemcitabine (Active Comparator)
  Interventions: Drug: Nab-paclitaxel Plus Gemcitabine
- Surufatinib with Nab-paclitaxel, and Gemcitabine (Other)
  Interventions: Drug: Surufatinib with Nab-paclitaxel, and Gemcitabine

INTERVENTIONS:
Drug: Surufatinib Combined With Camrelizumab, Nab-paclitaxel, and Gemcitabine — Drug: Surufatinib Combined With Camrelizumab, Nab-paclitaxel, and Gemcitabine
  1. Surufatinib: 200mg, qd
  2. Camrelizumab: 200mg, IV drip, Q3W, D1
  3. Nab-paclitaxel: 125 mg/m2, IV drip, D1,D8
  4. Gemcitabine : 1000 mg/m2, IV drip, D1, D8
  Arms: Surufatinib Combined With Camrelizumab, Nab-paclitaxel, and Gemcitabine
Drug: Nab-paclitaxel Plus Gemcitabine — Drug: Nab-paclitaxel Plus Gemcitabine
  1. Nab-paclitaxel: 125 mg/m2, IV drip, D1,D8
  2. Gemcitabine : 1000 mg/m2, IV drip, D1, D8
  Arms: Nab-paclitaxel Plus Gemcitabine
Drug: Surufatinib with Nab-paclitaxel, and Gemcitabine — Drug: Surufatinib with Nab-paclitaxel, and Gemcitabine
  1. Surufatinib: 200mg, qd
  2. Nab-paclitaxel: 125 mg/m2, IV drip, D1,D8
  3. Gemcitabine : 1000 mg/m2, IV drip, D1, D8
  Arms: Surufatinib with Nab-paclitaxel, and Gemcitabine

SUMMARY:
To evaluate the efficacy of surufatinib combined with camrelizumab, nab-paclitaxel, and gemcitabine versus nab-paclitaxel plus gemcitabine as the first-line treatment in metastatic pancreatic cancer

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active-controlled, phase II/III trial to evaluate the efficacy and safety of surufatinib combined with camrelizumab, nab-paclitaxel, and gemcitabine versus nab-paclitaxel plus gemcitabine as the first-line treatment in metastatic pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily sign an informed consent form, willing and able to follow the study process;
2. Age range is 18-75 years old (inclusive);
3. Pancreatic cancer confirmed by histology or cytology;
4. Stage IV metastasis Pancreatic cancer patients;
5. Have not received previous systematic first line anti-tumor treatment in the stage of metastatic pancreatic cancer;
6. According to RECIST 1.1, there is at least one measurable lesion;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1;
8. Expected survival time ≥ 12 weeks;

Exclusion Criteria:

1. Use of systematic anti-tumor therapy within 2weeks prior to the first dose；
2. Presence of other malignancies in the past 5 years;
3. Received major surgical surgery within 60 days before the first dose;
4. Have received any surgery or invasive treatment within 4 weeks before the first use of the drug;
5. Received palliative radiotherapy within 1 week before the first dose; received radical radiotherapy within 4 weeks before the first dose;
6. Any known allergy to surufatinib or its components, camrelizumab, nab-paclitaxel, or gemcitabine;
7. Received inducers or inhibitors of cytochrome P450 (CYP) 3A within 2 weeks or 5 half-lives (whichever is longer) before the first dose;
8. Use of immunosuppressive drugs within 4 weeks before first dose;
9. Known history of clinically significant liver disease, including active viral hepatitis infection or other active hepatitis or clinically significant moderate to severe cirrhosis;
10. Patients who currently have hypertension that cannot be controlled by medication;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of first dose of study drug until withdrawal of consent or death (up to approximately 20 months)
  Duration from the date of initial treatment to the date of death due to any cause

SECONDARY OUTCOMES:
Progression-free Survival (PFS) (RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy (up to approximately 20 months)
  A duration from the date of initial treatment to disease progression or death of any cause.
Objective response rate (ORR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy (up to approximately 20 months)
  The incidence of confirmed complete response or partial response
Duration of response (DoR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy (up to approximately 20 months)
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Disease control rate (DCR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy (up to approximately 20 months)
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30)（only for phase III） | From the within 7 days prior to the initiation of treatment to 30 days after the last administration
  The changes in health-related quality of life (HRQoL) score from baseline and the time to deterioration of symptoms (TTD) as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire
  - Core 30 (EORTC QLQ-C30)
Cancer Quality of Life Questionnaire - PAN26(EORTC QLQ-PAN26)（only for phase III） | From the within 7 days prior to the initiation of treatment to 30 days after the last administration
  The changes in health-related quality of life (HRQoL) score from baseline and thehe time to deterioration of symptoms (TTD) as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire
  - PAN26 (EORTC QLQ-PAN26)
Safety and tolerability | From the date of first dose of study drug to 90 days after the last administration
  Incidence and nature of treatment emergent adverse events(TEAE), the other safety variables including physical examination, vital signs and laboratory examinations.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing Tianyinshan Hospital, Nanjing, Jiangsu
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No